CLINICAL TRIAL: NCT03110731
Title: Effect of Strength Training on the Quality and Duration of Sleep and Daytime Sleepiness of Institutionalized Adolescents: A Randomized Study
Brief Title: Effect of Strength Training on the Quality and Duration of Sleep and Daytime Sleepiness of Institutionalized Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Responsible Party: Principal Investigator, Rodrigo Pinto Pedrosa, Director of Sleep and Heart Laboratory, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STRENGTH trial
Record Dates: First submitted 2017-04-01; First posted 2017-04-12 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Adolescent Behavior; Sleep Disorder
MeSH Terms: conditions — Adolescent Behavior; Sleep Wake Disorders | interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Physical training (2x / week) was performed for 12 weeks
  Interventions: Behavioral: Physical training
- Control Group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Physical training — Physical training (2x / week) was performed for 12 weeks
  Arms: Intervention group

SUMMARY:
The aim of this study was to analyze the effects of strength training on sleep quality and daytime sleepiness in institutionalized adolescents (14 to 19 years of age). Thirty-one adolescents were randomly assigned in two sample groups: intervention group (IG, n = 19) and control group (CG, n = 12). Anthropometric measures were performed (height and body mass) and BMI was determined. Sleep quality and daytime sleepiness were assessed using the questionnaires, Pittsburgh Sleep Quality Index (PSQI) and Epworth Sleepiness Scale (ESE), and total sleep time by accelerometer. Physical training (2x / week) was performed for 12 weeks. The OMNI Perceived Exertion Scale for Resistance Exercise (OMNI-RES) scale was used to control the effort intensity and the exercises followed an alternate pre-follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized adolescents (14 to 19 years of age)

Exclusion Criteria:

* refuse to participate,
* incomplete evaluation

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-24 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
sleep quality | 12 weeks
  improvement in Pittsburgh Sleep Quality Index (PSQI)
Daytime sleepiness | 12 weeks
  improvement Epworth Sleepiness Scale (ESE)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santiago LCS, Lyra MJ, Germano-Soares AH, Lins-Filho OL, Queiroz DR, Prazeres TMP, Mello MT, Pedrosa RP, Falcao APST, Santos MAM. Effects of Strength Training on Sleep Parameters of Adolescents: A Randomized Controlled Trial. J Strength Cond Res. 2022 May 1;36(5):1222-1227. doi: 10.1519/JSC.0000000000003629. Epub 2020 Apr 29. PMID 32379244